CLINICAL TRIAL: NCT06110949
Title: Thromboembolic Risk Assessment in Patients Admitted With Acute Medical Diseases to Conventional and At Home Hospitalization Units (TROMBODOM/ADOMFIB Study)
Brief Title: Thromboembolic Risk Assessment in Patients Admitted With Acute Medical Diseases to Conventional and At Home Hospitalization
Acronym: TROMBODOM
Status: Recruiting | Type: Observational
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Sociedad Española De Medicina Interna (Other); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: PI_2021/100//PI_2022/91
Record Dates: First submitted 2023-08-31; First posted 2023-11-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Thromboprophylaxis; Thromboembolism, Venous; Atrial Fibrillation; Physical Inactivity; Hospital at Home
Keywords: Thromboprophylaxis; Thromboembolism; Atrial Fibrillation; Accelerometry; Hospital at Home
MeSH Terms: conditions — Venous Thromboembolism; Atrial Fibrillation; Sedentary Behavior; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- At home hospitalization cohort: Participants admitted with acute medical diseases to at home hospitalization units will be included in a prospective registry in order to investigate the 90 days incidence of thromboembolic disease. A group of such patients will be controlled with triaxial accelerometer in order to collect raw data regarding patient mobility during admission.
  Interventions: Device: Triaxial accelerometry
- Conventional hospitalization cohort: Participants admitted with acute medical diseases to a conventional hospitalization unit will be included in a prospective registry in order to investigate the 90 days incidence of thromboembolic disease. A group of such patients will be controlled with triaxial accelerometer in order to collect raw data regarding patient mobility during admission.
  Interventions: Device: Triaxial accelerometry

INTERVENTIONS:
Device: Triaxial accelerometry — A group of patients will be controlled with triaxial accelerometer (GENEActiv watch) on left wrist at a sampling rate of 85,70 Hz to measure movement in the x, y, and z direction, in order to collect raw data regarding patient mobility (duration of sleep, the time spent in sedentary attitudes and the amount of light, moderate and vigorous physical activity) during the admission (from the admission day to discharge).

SUMMARY:
The thromboembolic disease is a common complication of patients admitted to conventional hospitalization units. To prevent such complications, thromboprophylaxis is indicated in high-risk patients identified with validated risk-assessment models such as Padua score and IMPROVE-VTE score. However, the relation between thromboembolic disease and inpatients is yet to be demonstrated in new clinical settings such as at home hospitalization units. Moreover, patient immobilization is key in the pathogenesis of thromboembolic complications: therefore, it is crucial to collect raw data of patient mobility during admission.

The goal of this observational study is to compare the thromboembolic risk of patients admitted with acute medical diseases to at home hospitalization units with conventional hospitalization units.

The main questions it aims to answer are:

* Is the estimated thromboembolic risk of patients admitted with acute medical diseases to at home hospitalization units similar to those admitted to conventional hospitalization units?
* Are the risk-assessment models used to predict thromboembolic risk of patients admitted with acute medical diseases to conventional hospitalization units (Padua and IMPROVE-VTE score) valid in at home hospitalization patients?

Participants admitted with acute medical diseases to either a conventional hospitalization unit or at home hospitalization units will be included in a prospective registry in order to investigate the 90 days incidence of thromboembolic disease. A cohort of such patients will be controlled with triaxial accelerometer in order to collect raw data regarding patient mobility during admission.

DETAILED DESCRIPTION:
1953 patients will be recruited (1700 in at home hospitalization units and 253 in conventional hospitalization units). All patients must accept and sign the informed consent. After being admitted to the study, patients will be included in the prospective registry with baseline evaluation of basic clinical data, including risk-assessment models (Padua and IMPROVE-VTE scores), examination, ECG, self-assessed mobility, and biochemistry markers. Triaxial accelerometers will also record mobility and sleep time of 135 patients from conventional hospitalization units and 135 patients from at home hospitalization units, from which physical activity questionnaires (International Physical Activity Questionnaire (IPAQ), The Spanish Short Version of the Minnesota Leisure Time Physical Activity Questionnaire (VREM)), handgrip strength, 30-second sit-to-stand test, the Short Physical Performance Battery (SPPB), the Spanish Version of 5-level European Quality of Life-5 Dimensions (5-level EQ-5D), Fried frailty criteria and Lobo's cognitive mini-examination will also be obtained. All 1953 patients will be followed for 90 days after discharge to assess thromboembolic disease incidence (pulmonary embolism, deep venous thrombosis, and atrial fibrillation), major and clinically relevant non-major bleedings (according to International Society on Thrombosis and Haemostasis Standards) and death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients admitted with acute medical diseases to either a conventional hospitalization unit or at home hospitalization units
* Capable and willing to provide an informed consent

Exclusion Criteria:

* End of life disease, palliative care or with an expected survival inferior to 3 months
* Patients receiving therapeutic doses of any anticoagulant drug
* Active diagnosis of thromboembolic disease
* Prior diagnosis of atrial fibrillation
* Pregnancy or breast-feeding.
* SARS-CoV-2 diagnosed using real-time reverse transcriptase polymerase chain reaction (PCR) tests or positive for SARS-CoV-2 virus antigen <90 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with acute medical diseases (non-surgical setting) to either a conventional hospitalization unit or at home hospitalization units, whenever able to understand the study protocol and sign the informed consent form, will be offered to participate in this study. In patients' best interests, those with end-of-life disease, receiving palliative care or with an expected life survival inferior to 3 months will not be included. To correctly evaluate the study outcomes, patients receiving therapeutic doses of any anticoagulant drug, those with active diagnosis of thromboembolic disease or prior diagnosis of atrial fibrillation will not be included. Finally, this study excludes pregnant or breast-feeding people and patients with active or recent SARS-CoV2 infection, due to well recognized differences in the pathophysiology of thromboembolic disease in such populations.
Sampling Method: Non-Probability Sample
Enrollment: 1953 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Estimated thrombotic risk at admission measured with Padua score | Within 3 months after hospitalization
  Estimated thrombotic risk of patients admitted with acute medical diseases to at home hospitalization units and conventional hospitalization units will be measured with Padua score (high or low risk). "Padua" score is a risk assessment model that scores from 0 to 20, with a score of 4 or higher identifying patients at "high risk" of thromboembolic disease.
Estimated thrombotic risk at admission measured with IMPROVE-VTE score | Within 3 months after hospitalization
  Estimated thrombotic risk of patients admitted with acute medical diseases to at home hospitalization units and conventional hospitalization units will be measured with IMPROVE-VTE score (high or low risk). "IMPROVE-VTE" score is a risk assessment model that scores from 0 to 12, with a score of 2 or higher identifying patients at "high risk" of thromboembolic disease.
Estimated hemorrhagic risk at admission | Within 3 months after hospitalization
  Estimated hemorrhagic risk of patients admitted with acute medical diseases to at home hospitalization units and conventional hospitalization units will be measured with IMPROVE-Bleeding score (high or low risk). "IMPROVE-Bleeding" score is a risk assessment model that scores from 0 to 33, with a score of 7 or higher identifying patients at "high risk" of hemorrhagic events.
Incidence of thrombotic events | Within 3 months after hospitalization
  Incidence of thrombotic events (deep venous thrombosis and pulmonary embolism) of patients admitted with acute medical diseases to at home hospitalization units and conventional hospitalization units
Incidence of atrial fibrillation diagnosis | Within 3 months after hospitalization
  Incidence of atrial fibrillation diagnosis in patients admitted with acute medical diseases to at home hospitalization units and conventional hospitalization units
Accelerometry | The duration of the hospitalization, from 0,9 days to 9 days
  A GENEActiv watch will be used on left wrist at a sampling rate of 85,70 Hz to measure movement in the x, y, and z direction. The results will be the duration of sleep, the time spent in sedentary attitudes and the amount of light, moderate and vigorous physical activity. All the outcomes may range from 1 to 1440 minutes per day.

SECONDARY OUTCOMES:
Prevalence of reduced mobility, measured with self-perceived immobilization | Baseline
  Self-perceived immobilization evaluated at admission with Padua score. "Padua" score is a risk assessment model that scores from 0 to 20, with a score of 4 or higher identifying patients at "high risk" of thromboembolic disease, and in which "reduced mobility" scores 3 points.
Prevalence of reduced mobility, measured with accelerometry | The duration of the hospitalization, from 0,9 days to 9 days
  Reduced mobility will be assessed in an objective determination with a GENEActiv watch. A GENEActive watch will be used on left wrist at a sampling rate of 85,70 Hz to measure movement in the x, y, and z direction. The results will be the duration of sleep, the time spent in sedentary attitudes and the amount of light, moderate and vigorous physical activity. All the outcomes may range from 1 to 1440 minutes per day.
Concordance of self-perceived immobilization and objective accelerometry measurements of physical activity for reduced mobility identification | At admission and during the duration of the hospitalization, from 0,9 days to 9 days
  Reduced mobility can be assessed by subjective (e.g. self-perceived immobilization) or objective means (accelerometry). This outcome will determine the variability in identifying reduced mobility patients, when comparing reduced mobility assessed by subjective (self-perceived immobilization) or objective means (accelerometry)
International Physical Activity Questionnaire (IPAQ) | First day of hospitalization and 3 months after hospitalization
  The IPAQ is a validated 7-day recall questionnaire measuring current levels of physical activity. This questionnaire will be administered to participants aged under 65 years old. Scoring of the IPAQ results in a continuous variable in the form of total METs per week, which may be converted to METs per day. Higher scores means higher physical activity level. Additionally, walking, moderate physical activity and intense physical activity will be calculated as minutes per week. In addition, we will measure the change in physical activity levels from before hospitalization to three months later.
The Spanish Short Version of the Minnesota Leisure Time Physical Activity Questionnaire (VREM) | First day of hospitalization and 3 months after hospitalization
  The VREM is a 6-item questionnaire that measures leisure time physical activity. It will be administered to people over 65 years of age. It reports energy expenditure over the past month expressed as 14-day METs. The number of METs per day will also be indicated. In addition, we will measure the change in physical activity levels from before hospitalization to three months later.
Handgrip strength | First (baseline) and last day of hospitalization (up to 9 days)
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.
30-second sit-to-stand test | First (baseline) and last day of hospitalization (up to 9 days)
  Participants under 65 years of age will repeat as many of the sit-to-stand actions as possible in 30 seconds and the maximum number completed will be recorded.
The Short Physical Performance Battery (SPPB) | First (baseline) and last day of hospitalization (up to 9 days)
  Participants over the age of 65 will complete the SPPB, which consists of 3 tests: 1) a progressive test of standing balance, 2) a 4-meter usual pace walk, and 3) a five-repetition chair stand test. Each test has a minimum score of 0 points and a maximum of 4 points. Thus, the final SPPB score ranges from 0 to 12 points.
The Spanish Version of 5-level European Quality of Life-5 Dimensions (5-level EQ-5D) | First day of hospitalization (baseline)
  The 5-level EQ-5D (EQ-5D-5L) is a generic standardized instrument that will be used to describe and assess the health-related quality of life of people over 65 years of age. The 5-level EQ-5D (EQ-5D-5L) instrument consists of two parts: the EQ-5D descriptive system and the Visual Analogue Scale (VAS). The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. In the VAS, the individual scores his or her health between two extremes, 0 being the worst imaginable state of health and 100 the best imaginable state of health.
Fried frailty criteria | First day of hospitalization (baseline)
  Frailty in people older than 65 years will be assessed according to five criteria: unintentional weight loss, low mood, gait speed, level of physical activity and muscle weakness. The stages of frailty have been defined as follows: a score of 0 means that a person is robust or not frail, a score of 1 or 2 indicates a risk for adverse outcomes and is considered to pre-frailty and a score of 3-5 suggests that the person is frail.
Lobo's cognitive mini-examination | First day of hospitalization (baseline)
  This questionnaire examines several cognitive dimensions: temporal orientation, spatial orientation, attention, concentration and calculation, memory and language and construction. In people over 65 years of age, scores of 23-24 are the cut-off point at which a diagnosis of dementia is established. A score between 20 and 24 indicates mild cognitive impairment. Values between 15 and 19 represent moderate cognitive impairment and a clear sign of the existence of dementia. Finally, a score below 15 points suggests severe cognitive impairment leading to advanced dementia.
Prevalence of pharmacological thromboprophylaxis use | Last day of hospitalization (up to 9 days)
  Prevalence of pharmacological thromboprophylaxis (low molecular weight heparin) use during admission
Prevalence of correct pharmacological thromboprophylaxis use according to risk assessment models | Last day of hospitalization (up to 9 days)
  Prevalence of correct pharmacological thromboprophylaxis (low molecular weight heparin) use during admission, evaluated according to Padua and IMPROVE-VTE score
Prevalence of correct pharmacological thromboprophylaxis use according to objective mobility evaluation with accelerometry | Last day of hospitalization (up to 9 days)
  Prevalence of correct pharmacological thromboprophylaxis (low molecular weight heparin) use during admission, evaluated according to Padua and IMPROVE-VTE score when mobility is evaluated objectively with accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Joao Modesto dos Santos, Medical Doctor, Principal Investigator — Hospital Universitario de Navarra, Spain
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No